CLINICAL TRIAL: NCT00376844
Title: PORTEC-2, Postoperative Radiation Therapy for Endometrial Carcinoma - A Multicenter Randomised Phase III Trial Comparing External Beam Radiation and Vaginal Brachytherapy
Brief Title: External-Beam Radiation Therapy Compared With Vaginal Brachytherapy After Surgery for Stage I Endometrial Cancer
Acronym: PORTEC-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Carien Creutzberg, Professor of Radiation Oncology, Chief investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000502033; CKTO-2001-04 (Other Grant/Funding Number: Dutch Cancer Society); P01.146 (Other: LUMC Ethics Committee); ISRCTN16228756 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Intervention Model Description: Exterbal beam radiation therapy versus vaginal brachytherapy
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Beam Radiation Therapy (Active Comparator): Postoperative pelvic radiotherapy
  Interventions: Radiation: External Beam Radiation Therapy
- Vaginal Brachytherapy (Experimental): Postoperative vaginal brachytherapy
  Interventions: Radiation: Vaginal Brachytherapy

INTERVENTIONS:
Radiation: External Beam Radiation Therapy
  Other Names: pelvic radiotherapy
  Arms: External Beam Radiation Therapy
Radiation: Vaginal Brachytherapy
  Other Names: internal radiation
  Arms: Vaginal Brachytherapy

SUMMARY:
RATIONALE: External-beam radiation therapy uses high-energy x-rays to kill tumor cells. Implant radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving external-beam radiation therapy or implant radiation therapy after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether radiation therapy is more effective than observation when given after surgery in treating stage I endometrial cancer.

PURPOSE: This randomized phase III trial is studying external-beam radiation therapy or implant radiation therapy to see how well they work compared with observation in treating patients who have undergone surgery for stage I endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rate of 5-year locoregional relapse in patients undergoing external-beam radiotherapy or vaginal brachytherapy vs observation only after surgery for stage I endometrial cancer.
* Compare 5-year rate of distant metastases in these patients.
* Determine overall survival rate in these patients.
* Determine prognostic factors for relapse and morbidity.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo either vaginal brachytherapy or external-beam radiotherapy.
* Arm II: Patients are observed and undergo no further treatment. After completion of study treatment, patients are followed for approximately 83 days.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of FIGO 1988 stage I-IIA endometrial cancer, meeting 1 of the following criteria:

  * Age ≥60, stage IC grade 1 or 2 with deep (≥ 50%) myometrial invasion
  * Age ≥60, stage IB grade 2 or 3 (with < 50% myometrial invasion)
  * Stage IIA, any age
* No grade 3 endometrial carcinoma with deep myometrial invasion
* Total abdominal hysterectomy and bilateral salpingo-oophorectomy required prior to randomisation
* WHO performance status 0-2

EXCLUSION CRITERIA:

* Serous or clear cell histology or uterine sarcoma
* staging lymphadenectomy
* interval between surgery and radiotherapy > 8 weeks
* history of previous malignant disease (except basal cell carcinoma of skin)
* previous radiotherapy, hormonal therapy or chemotherapy
* diagnosis of Chrohn's disease or ulcerative colitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2002-05; Primary Completion 2009-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Vaginal relapse | 5 years
  total vaginal relapse and vaginal relapse as first failure

SECONDARY OUTCOMES:
Rate of distant metastases | 5 years
  total distant relapse and distant relapse as first failure
Overall survival | 5 years
  all-cause survival (and cancer-related survival)
Adverse effects | 5 years
  Types and severity graded according to EORTC-RTOG grading system
Health-related quality of life | 5 years
  Cancer-specific quality of life (EORTC QLQ C-30); patient reported symptoms
Pelvic relapse | 5 years
  total pelvic relapse and pelvic relapse as first failure

CONTACTS AND LOCATIONS:
Overall Officials: Carien L. Creutzberg, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After submission of a research plan and approval by the TMG data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] McCloskey SA, Tchabo NE, Malhotra HK, Odunsi K, Rodabaugh K, Singhal P, Lele S, Jaggernauth W. Adjuvant vaginal brachytherapy alone for high risk localized endometrial cancer as defined by the three major randomized trials of adjuvant pelvic radiation. Gynecol Oncol. 2010 Mar;116(3):404-7. doi: 10.1016/j.ygyno.2009.06.027. Epub 2009 Nov 27. PMID 19944453
- [Result] Nout RA, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Stenfert Kroese MC, Nijman HW, van de Poll-Franse LV, Creutzberg CL. Five-year quality of life of endometrial cancer patients treated in the randomised Post Operative Radiation Therapy in Endometrial Cancer (PORTEC-2) trial and comparison with norm data. Eur J Cancer. 2012 Jul;48(11):1638-48. doi: 10.1016/j.ejca.2011.11.014. Epub 2011 Dec 14. PMID 22176868
- [Result] Nout RA, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Stenfert Kroese MC, van Bunningen BN, Smit VT, Nijman HW, van den Tol PP, Creutzberg CL. Quality of life after pelvic radiotherapy or vaginal brachytherapy for endometrial cancer: first results of the randomized PORTEC-2 trial. J Clin Oncol. 2009 Jul 20;27(21):3547-56. doi: 10.1200/JCO.2008.20.2424. Epub 2009 Jun 22. PMID 19546404
- [Result] Nout RA, Putter H, Jürgenliemk-Schulz IM, et al.: Vaginal brachytherapy versus external beam pelvic radiotherapy for high-intermediate risk endometrial cancer: Results of the randomized PORTEC-2 trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-LBA5503, 2008.
- [Result] Nout RA, Smit VT, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Kroese MC, van Bunningen BN, Ansink AC, van Putten WL, Creutzberg CL; PORTEC Study Group. Vaginal brachytherapy versus pelvic external beam radiotherapy for patients with endometrial cancer of high-intermediate risk (PORTEC-2): an open-label, non-inferiority, randomised trial. Lancet. 2010 Mar 6;375(9717):816-23. doi: 10.1016/S0140-6736(09)62163-2. PMID 20206777
- [Result] de Boer SM, Nout RA, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Stenfert Kroese MC, Oerlemans S, Putter H, Verhoeven-Adema KW, Nijman HW, Creutzberg CL. Long-Term Impact of Endometrial Cancer Diagnosis and Treatment on Health-Related Quality of Life and Cancer Survivorship: Results From the Randomized PORTEC-2 Trial. Int J Radiat Oncol Biol Phys. 2015 Nov 15;93(4):797-809. doi: 10.1016/j.ijrobp.2015.08.023. Epub 2015 Aug 18. PMID 26530748
- [Derived] Horeweg N, Nout RA, Jurgenliemk-Schulz IM, Lutgens LCHW, Jobsen JJ, Haverkort MAD, Mens JWM, Slot A, Wortman BG, de Boer SM, Stelloo E, Verhoeven-Adema KW, Putter H, Smit VTHBM, Bosse T, Creutzberg CL; PORTEC Study Group. Molecular Classification Predicts Response to Radiotherapy in the Randomized PORTEC-1 and PORTEC-2 Trials for Early-Stage Endometrioid Endometrial Cancer. J Clin Oncol. 2023 Sep 20;41(27):4369-4380. doi: 10.1200/JCO.23.00062. Epub 2023 Jul 24. PMID 37487144
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.clinicaltrials.gov/ct2/show/study/NCT00376844?term=portec&cond=Endometrial+Cancer&rank=1